CLINICAL TRIAL: NCT05912270
Title: Orchestra in Class, a Novel Booster for Executive Functions and Brain Development in Young Primary School Children
Acronym: ORBIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Collaborators: University of Geneva, Switzerland (Other); University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Clara E James, Full Professor HES-SO, School of Health Sciences Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 126645
Record Dates: First submitted 2023-05-30; First posted 2023-06-22 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Development, Child; Executive Functions; Interventions; Music; Arts; Brain Plasticity; Behavior; Brain Imaging; Magnetic Resonance Imaging; Functional Magnetic Resonance Imaging; Structural Brain Connectivity
MeSH Terms: conditions — Arts syndrome; Behavior | interventions — Artifacts

STUDY DESIGN:
Intervention Model Description: The study is a 1) block-randomized, 2) 3-arm, 3) open, 4) monocentric (primary schools in Geneva) 5) national (Switzerland) 6) intervention study.
Who Masked: Participant
Masking Description: Orchestra in Class is the first Experimental Condition, compared to Visual Arts (second Experimental Condition) and an active Control Group that will receive 6 cultural outings per year. We will present the study to the participants as a comparison between the two art interventions and a cultural intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Orchestra in Class (Experimental): Children will receive music practice lessons in groups, "Orchestra in Class" (4 different string instruments, violin, viola, cello, double bass) in school class size groups over 2 full years. Interventions, given by 2 professional teachers per class, take place for 1 hour and 30 minutes per week, completed by daily homework (20-30 minutes).
  Interventions: Behavioral: Orchestra in Class
- Visual Arts (Experimental): Children will receive visual arts lessons in school class size groups over 2 full years. Interventions, given by 2 professional teachers per class, take place for 1 hour and 30 minutes per week, completed by daily homework (20-30 minutes).
  Interventions: Behavioral: Orchestra in Class
- Culture (Placebo Comparator): The children will receive six cultural outings per year (museums, concerts, theatre, etc.) and pass all measurements
  Interventions: Behavioral: Orchestra in Class

INTERVENTIONS:
Behavioral: Orchestra in Class — See arm/group descriptions
  Other Names: Visual Arts

SUMMARY:
How to optimally stimulate the developing brain is still unclear. Executive functions (EF) exhibited substantially stronger far transfer effects in children who learned to play a musical instrument than in children who acquired other arts.

What is crucially lacking is a large-scale, long-term genuine randomized controlled trial (RCT) in cognitive neuroscience, comparing musical instrumental training (MIP) to another art form and a control group. Collected data of this proposal will allow, using machine learning, to build a data-driven multivariate model of children's interconnected brain and EF development over the first 2 years of their academic curriculum (6-8 years), with or without music or other art training.

DETAILED DESCRIPTION:
This cognitive neuroscience study, employing a randomized controlled trial (RCT), aims to investigate the potential cognitive and brain development benefits in young school children from two-year interventions: Orchestra in Class (OC, music practice, experimental group) compared with Visual Arts (VA, second experimental group) versus Standard Education (active control group (CG)). The CG will be offered six cultural outings per year (concerts, museums, theatres, etc.). Both nonverbal art interventions will be given weekly interventions for 1 hour and 30 minutes in school class sized groups. The VA groups serve to control for the influences of regular stimulating group interventions and homework, and also to compare specific effects in visual mode with the auditory mode in OC. The CG controls for overall child development and test-retest effects.

We plan to recruit 150 children aged 6-8 years from public elementary schools, ensuring a random and therefore equal distribution among the three groups. Data collection will involve annual comprehensive psychometric testing (baseline, after 1 year, after 2 years) of executive functions, i.e., far transfer and near transfer, musicality, drawing, academic achievement, and multimodal structural and functional magnetic resonance imaging (fMRI), including fMRI with auditory and visual domain working memory tasks.

By utilizing multivariate analyses and integrating behavioral and brain data through machine learning, we aim to create a data-driven model of the development of executive functions at the behavioral and brain levels in young children at the beginning of their school careers (6 to 8 years old), both without and with an enriched environment (musical practice versus visual arts)

ELIGIBILITY:
Inclusion Criteria:

* School grade 3P/4P (3rd and 4th year of elementary school (6-8-year-old children)
* Right-handedness
* Sufficient Mastery of the French Language
* Able to give oral informed consent (child)
* Able to give written informed consent (parent)

Exclusion Criteria:

* Non-consent (children and or parents)
* Repeated or skipped a class with respect to standard curriculum
* Not corrected/severe hearing deficits
* Not corrected/severe vision deficits
* Severe neurodevelopmental disorders (eg. severe dyslexia, severe ADHD)
* Older than 7 at the beginning of the school year if 3P
* Older than 8 at the beginning of the school year if 4P
* Protocolled music instrumental practice in the preceding year
* Protocolled visual arts courses in the preceding year
* MRI incompatibility (physical or psychological)
* Psychometric battery incompatibility (psychological)

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-12-18 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Working Memory | 2 years
  Working memory (WM) will be assessed by 3 tests: 2 fMRI tests: a visual and an auditory WM test (Vuontela et al., 2003) and the Digit Span Backward from the WISC V (Wechsler Intelligence Scale for Children; Wechsler, 2014).
  We expect the progress of the mean WM score to show the following evolution after 2 years:
  Orchestra in Class > Visual Arts > Passive Control Group

SECONDARY OUTCOMES:
Plasticity of gray matter brain volume | 2 years
  Gray matter brain plasticity, measured by T1-weighted MRI MP2RAGE (magnetization prepared 2 rapid acquisition gradient echoes; Marques & Gruetter, 2013)
  We expect greater gray matter volume change after 2 years according to the following gradient:
  Orchestra in Class > Visual Arts > Passive Control Group
  For the following brain areas:
  notably in a set of temporal (medial and lateral (auditory)), prefrontal, superior parietal areas, the basal ganglia (striatum), the cerebellum and the corpus callosum (supporting Working Memory, Executive Functions and attention)
Functional brain connectivity | 2 years
  Functional brain connectivity, measured with resting-state functional MRI (Leonardi,et al., 2013)
  We anticipate greater Functional Connectivity (FC) changes following the same gradient
  Orchestra in Class > Visual Arts > Passive Control Group
  In the following brain networks:
  The Default Mode Network (DMN), Central Executive Network (CEN) and Salience Network (SN)

CONTACTS AND LOCATIONS:
Overall Officials: Clara James, PhD, Study Director — HES-SO University of Applied Sciences and Arts Western Switzerland
Locations (1):
- Haute école de santé de Genève HES-SO, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No
At the end of the project, the recoded data set (cleaned and anonymized excel and R file formats, matlab matrices, all scripts), the data codebook, references for the measurement instruments and all other relevant information related to the project (protocol, sampling, etc.) will be deposited at the Yareta (DLCM Data Life Cycle Management) platform for data sharing and reuse. Potential users will be informed of data availability by means of explicit mentions in publications (e.g., section "availability of data and material" in publications). The contact and identity information of the participants will never be shared.

REFERENCES:
- [Derived] James CE, Tingaud M, Laera G, Guedj C, Zuber S, Diambrini Palazzi R, Vukovic S, Richiardi J, Kliegel M, Marie D. Cognitive enrichment through art: a randomized controlled trial on the effect of music or visual arts group practice on cognitive and brain development of young children. BMC Complement Med Ther. 2024 Apr 4;24(1):141. doi: 10.1186/s12906-024-04433-1. PMID 38575952